CLINICAL TRIAL: NCT01618097
Title: Evaluation of DVD and Internet Decision Aids for Hip and Knee Osteoarthritis: Focus on Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00032794
Record Dates: First submitted 2012-05-29; First posted 2012-06-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Decision Aids; Health Literacy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVD Decision Aid (Experimental): Patient assigned to watch DVD decision aid.
  Interventions: Behavioral: DVD Decision Aid
- Internet Based Decision Aid (Experimental): Patient assigned to watch OA specific internet based decision aid.
  Interventions: Behavioral: Internet Based Decision Aid

INTERVENTIONS:
Behavioral: DVD Decision Aid — Patients will receive the DVD decision aid to view, and follow up 3 days and 30 days post visit.
  Arms: DVD Decision Aid
Behavioral: Internet Based Decision Aid — Patients will receive the OA specific internet based decision aid to view, and follow up 3 days and 30 days post visit
  Arms: Internet Based Decision Aid

SUMMARY:
The purpose of this study is to advance the evidence base regarding methods for facilitating informed decisions among patients with knee and hip osteoarthritis by comparing DVD and online formats of decision aids for these conditions. The project will assess how these different formats impact key outcomes including: patient knowledge about treatment options, decisional conflict, preparation for decision making, decision self-efficacy, stage of decision making, and acceptability and usability of the decision aids.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common chronic conditions and a leading cause of pain and disability. Many patients with OA know very little about treatment options and are not well equipped to make informed decisions regarding these treatments. Further, there are racial and gender disparities in perceptions of the risks and benefits of total joint replacement, which also highlights the need to improve facilitation of informed treatment choices in these patients. Decision aids have great potential to improve patient satisfaction, safety, and outcomes for patients with OA, but there is no evidence base regarding best formats for delivering this information. This project will compare patient decision-making outcomes immediately following viewing of DVD and web-based versions of the Health Dialog DAs for hip and knee OA, as well as three days and one month later. Patients with symptomatic knee and hip OA (n=200) will be enrolled from a primary care and orthopedic clinics. Participants will be randomized, with stratification according to health literacy level, to view the DVD or web-based DA. Outcomes will include: Knowledge about OA and Treatments, Decisional Conflict, Preparation for Decision-Making, Decision Self-Efficacy, Stage of Decision Making, Acceptability and Usability of the DA, and home use of the DA. This project will make a novel contribution with direct clinical applicability, providing information regarding best methods for disseminating tools to enhance informed decision-making among patients with hip and knee OA, with particular attention to patients with low literacy.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of knee/hip OA, based on radiographic evidence in Duke medical records.
* Moderate or worse current joint symptoms, assessed at telephone screening using standard items.

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease.
* Active diagnosis of psychosis or dementia, or other cognitive impairment.
* Severe hearing or visual impairment that would prohibit effective use of the DAs.
* Planning, scheduled for or on a wait list for joint replacement surgery.
* Had a prior hip or knee joint replacement surgery.
* Inability to read English, since the DAs are in English.
* Current participation in another OA interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in the Facts about Osteoarthritis section of the Decision Quality Instrument - Knee Osteoarthritis (DQI-KOA; © Massachusetts General Hospital, 2010 46) at Baseline to post. | Baseline and 1 hour
  Knowledge is a key outcome in this study because it is fundamental to informed decision making process 45. We will use the "Facts about Osteoarthritis" section of the Decision Quality Instrument - Knee Osteoarthritis (DQI-KOA; © Massachusetts General Hospital, 2010 46), which includes 8 items that assess knowledge about the knee OA and its treatment options (behavioral, pharmacological, and surgical). Although this instrument was developed for knee OA, the items are also appropriate for hip OA, and it will be used for both groups.
Change in Decisional Conflict Scale at Baseline to post. | Baseline and 1 hour
  We will use the Low Literacy version of this scale, which includes 10 items with 3 response categories (yes, no, unsure), across four subscales: Informed (do patients know the different options, benefits, and risks?), Values Clarity (are patients clear about which benefits and risk matter most to them?), Support (do patients have support and advice to make a choice?), and Uncertainty (are patients clear or sure about what to choose?).
Change in Decision Self-Efficacy Scale a Baseline to post. | Baseline and 1 hour
  This is an 11-item scale that measures patients' confidence in completing various tasks related to the decision-making processes, such as getting facts about risks and benefits, asking questions, and expressing concerns. All items are measured on a scale of 0 (not confident at all) to 4 (very confident).
Change in the Facts about Osteoarthritis section of the Decision Quality Instrument - Knee Osteoarthritis (DQI-KOA; © Massachusetts General Hospital, 2010 46) at 30 days. | Baseline and 30 days
Change in Decisional Conflict Scale at 30 days post. | Baseline and 30 days

SECONDARY OUTCOMES:
Measurement of the Acceptability and Usability Scale post viewing of the DAs. | Up to 1 hour
  We will adapt a 10-item scale to assess the acceptability of this OA DAs. This tool assesses patients' opinions of general aspects of the DA (e.g., amount of information, length), as well as specific topical areas of the DA. In addition, for participants who are randomized to view the internet-based DA, we will use the Perceived Health Website Usability Questionnaire. This questionnaire includes items that assess the ease of finding information, ease of reading, appearance, and ease of learning from the website.
Semi-Structured Interviews | Up to 1 hour
  We will use semi-structured interviews to assess patients' perceptions and opinions of the DAs. Specific questions will be developed by the study team, covering the following topical areas: What participants liked about the DA, how well it answered questions they had about treatment options, any additional information to inform their decision-making, other suggestions for improving the DA, likelihood of using the DA to obtain information about treatment options, and how beneficial they think it would be to talk with a nurse / health educator about this information after viewing the DA.
Time spent viewing different parts of the internet-based DA | Up to 1 hour
  Installation of Spector Pro software onto the laptop computer on which participants will view the DA to capture information about participants' viewing of the DA. Descriptive data will be generated. Main variables we plan to evaluate are: 1.) The proportion of patients who view each page of the website. 2.) The mean or median number of minutes patients spent on each page. 3.) The proportion of patients who view video(s) within the DA. We will also compare these variables according to patient characteristics and changes in study outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Result] Allen, K.D., Sanders, L. Olsen, M., Bowlby, L., Katz, J.N., Mather, R.C., Powers, B., Sperber, N., Voils, C.I., Williams, J.W. Effectiveness of Internet and DVD Decision Aids for Patients with Hip and Knee Osteoarthritis. April 2014 World Congress on Osteoarthritis. Paris, France.